CLINICAL TRIAL: NCT01255137
Title: Phase II Study of Axitinib (AG-013736) With Evaluation of the VEGF-Pathway in Metastatic, Recurrent or Primary Unresectable Adrenocortical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100203; 10-C-0203
Record Dates: First submitted 2010-12-04; First posted 2010-12-07 (Estimated); Results first posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-04

CONDITIONS: Adrenal Cortex Neoplasms
Keywords: Selective VEGF Inhibitor; Clinical Activity; Response Rate; Measurable Disease; Biological Markers; Adrenocortical Cancer
MeSH Terms: conditions — Adrenal Cortex Neoplasms | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adrenal Cortex Neoplasms (Experimental): Aggressive cancer that starts in the adrenal gland located at the top of the kidneys.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — 5 mg tab orally twice a day with food every 28 days
  Other Names: AG-013736

SUMMARY:
Background:

- Adrenocortical carcinoma is an aggressive cancer that starts in the adrenal gland at the top of the kidneys. It has a low survival rate if standard treatment options are not effective. Axitinib is an experimental drug that is being studied to determine if it can stop tumors from growing or make them smaller. Researchers are interested in investigating axitinib in individuals with aggressive or otherwise untreatable adrenocortical cancer.

Objectives:

- To evaluate the effectiveness of axitinib in individuals who have adrenocortical cancer that is inoperable and has not responded to standard treatments.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with adrenocortical cancer that has not responded to standard treatments.

Design:

* Participants will be screened with a full physical examination and medical history, as well as tumor imaging studies.
* Participants may have a tumor biopsy prior to starting axitinib.
* All participants will receive axitinib to take twice a day with food for 28 days (1 cycle). Participants should not drink grapefruit juice or smoke cigarettes while participating in this study.
* After the first cycle, the dose may be increased and additional cycles will be given if the treatment has not had serious side effects.
* Participants will have regular examinations while taking axitinib, including blood samples and tumor imaging studies to determine if the tumor has stopped growing. Blood pressure levels will be carefully monitored during treatment to evaluate potential risk for high blood pressure.
* Participants may have a second tumor biopsy 20 to 30 days after treatment begins.
* Treatment will continue as directed by the study researchers.

DETAILED DESCRIPTION:
Background:

* The response rates of recurrent, metastatic and unresectable adrenocortical cancer (ACC) to mitotane, doxorubicin, etoposide, and cisplatin are low and underscore the need for more effective systemic therapies.
* VEGF expression and evidence of angiogenesis has been found in many ACCs, so it is plausible that interfering with vascular endothelial growth factor(VEGF) signaling may result in anti-tumor activity in patients with ACC.
* Axitinib (AG-013736) is an oral, potent and selective inhibitor of vascular endothelial growth factor (VEGF) receptors 1, 2, and 3. Pre-clinical data suggests that the anti-tumor activity of axitinib may result from its anti-angiogenic activity and that this is reversible when treatment is discontinued.
* Given the known clinical safety and efficacy of axitinib, an assessment of its activity in ACC and its impact on the VEGF pathway in ACC could provide valuable information.

Objectives:

* Determine the response rate of axitinib (AG-013736) in recurrent, metastatic, or primary unresectable ACC
* Determine the progression-free survival
* Explore the relationship of potential biological markers of axitinib activity with clinical outcomes.
* Explore the pharmacogenetic analyses of drug metabolism and transport proteins through germline deoxyribonucleic acid (DNA) examination.

Eligibility:

* Adults with pathologic confirmation of ACC by the Laboratory of Pathology, National Cancer Institute (NCI)
* Diagnosis of recurrent, metastatic, or primary unresectable ACC
* Measurable disease at presentation
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Patients must not have received prior therapy with a tyrosine kinase (TK) inhibitor

Design:

* Phase II, open label, non-randomized trial
* Patients with recurrent, metastatic, or primary unresectable ACC will be given in eight weeks cycles with BID dosing of axitinib (AG-013736).
* Patients will be evaluated for response every eight weeks using Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Tumor biopsies are not mandatory but every attempt will be made to obtain these from patients prior to starting axitinib and again 20-30 days after treatment has begun.
* Approximately 40 patients will be needed to achieve the objectives of the trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Pathologic confirmation of adrenocortical cancer by the Laboratory of Pathology, National Cancer Institute (NCI).
  2. Measurable disease at presentation.
  3. A life expectancy of at least 3 months and Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
  4. Age greater than or equal to 18 years.
  5. Last dose of chemotherapy or experimental therapy more than 4 weeks (6 weeks in the case of nitrosourea) prior to enrollment date; 2 weeks if the last therapy was received as part of a phase 0 or exploratory investigational new drug (IND) trial. Last surgery more than 4 weeks prior to enrollment, to allow for wound healing. Core biopsies or fine needle aspiration (FNA) will not require any waiting period.
  6. Last radiotherapy treatment 4 weeks prior to starting treatment with this protocol and there must be sites of measurable disease that did not receive radiation.
  7. Prior mitotane therapy is allowed. Patients with a history of a functional tumor who are receiving mitotane to control the excess hormone production may continue to receive mitotane.
  8. Organ and marrow function as defined below:
* Total bilirubin less than or equal to 1.5 x ULN (upper limit of normal), unless the patient meets the criteria for Gilbert's Syndrome. The upper limit value for bilirubin for subjects with Gilbert's Syndrome is less than 3 mg/dl.

Note: A diagnosis of Gilbert's disease will be made in the presence of (1) unconjugated hyperbilirubinemia noted on several occasions; (2) normal results from complete blood count (CBC) count, reticulocyte count, and blood smear; (3) normal liver function test results; and (4) an absence of other disease processes that can explain the unconjugated hyperbilirubinemia.

* Aspartate aminotransaminase (AST) less than or equal to 2.5 times ULN, alanine aminotransaminase (ALT) greater than or equal to 2.5 times ULN
* Amylase and lipase equal to, or less than, the institutional ULN.
* Creatinine clearance greater than or equal to 40 ml/min (measured in a timed urine collection) or serum creatinine less than or equal to 1.6 mg/dl
* Absolute neutrophil count greater than or equal to 1000/mm^3.
* Platelet count greater than or equal to 100,000/ mm^3.

  9. Ability to understand and sign an informed consent document.

  10. Ability and willingness to follow the guidelines of the clinical protocol including visits to NCI, Bethesda, Maryland for treatment and follow up visits.

  11. Because the effects of chemotherapy on the developing human fetus are potentially harmful, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier methods) before, during the study and for a period of 3 months after the last dose of chemotherapy.

EXCLUSION CRITERIA:

1. Patients with adrenocortical tumors potentially curable by surgical excision alone as determined by the Principal Investigator in discussions with the surgical consultants.
2. Patients who have large abdominal masses impinging on bowel or pulmonary masses with encroached vessels and a potential to bleed will be considered on case by case basis after careful consultation with multiple disciplines such as radiologists and surgeons with main intent being patient safety.
3. Unstable hypertension defined as a systolic blood pressure greater than 140 mm Hg or diastolic pressure greater than 90 mmHg despite optimal medical management and patients who are receiving more than 1 antihypertensive agent at trial entry, (not including spironolactone) unless the patient has Cushing's Disease with its associated hypertension and is well controlled on medications.
4. Untreated brain metastases (or local treatment of brain metastases within the last 6 months) due to the poor prognosis of these patients and difficulty ascertaining the cause of neurologic adverse events.
5. Pregnancy, due to the possible adverse effects on the developing fetus.
6. Lactating women who are breast-feeding due to the possibility of transmitting axitinib to the child.
7. The presence of a second malignancy, other than a skin cancer or in situ cervical cancer because it will complicate the primary objective of the study. Cancer survivors who have been free of disease for at least two years can be enrolled in this study.
8. Patients with evidence of a bleeding diathesis.
9. Phosphorus level equal to, or less than, the institutional lower limits of normal that cannot be corrected.
10. Gastrointestinal abnormalities including:

    1. inability to take oral medications
    2. requirement for intravenous alimentation
    3. prior surgical procedure affecting absorption including total gastric resection
    4. treatment for active peptic ulcer disease in the past 6 months
    5. active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy
    6. malabsorption syndrome
11. Current use or anticipated need for treatment with drugs that are known potent cytochrome P450 3A4 (CYP3A4) inhibitors (i.e., grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir, and delavirdine).
12. Current use or anticipated need for treatment with drugs that are known CYP3A4 inducers (i.e., carbamazepine, Phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampin, and St. John's wort).
13. Requirement of anticoagulant therapy with oral vitamin K antagonists. Low-dose anticoagulants for maintenance of patency of central venous access devise or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.
14. Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis.
15. Any of the following within 12 months prior to study drug administration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack and 6 months for deep vein thrombosis or pulmonary embolism.
16. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
17. Current use of drugs that are known inhibitors or inducers of Breast Cancer Resistance Protein (BCRP) and Organic Anion Transporting Polypeptide (OATP)1B1/3 or known to affect protein binding should be used with caution and with acknowledgement of the principal investigator (PI).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio T Fojo, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Plager JE. Carcinoma of the adrenal cortex: clinical description, diagnosis, and treatment. Int Adv Surg Oncol. 1984;7:329-53. No abstract available. PMID 6088397
- [Background] Luton JP, Cerdas S, Billaud L, Thomas G, Guilhaume B, Bertagna X, Laudat MH, Louvel A, Chapuis Y, Blondeau P, et al. Clinical features of adrenocortical carcinoma, prognostic factors, and the effect of mitotane therapy. N Engl J Med. 1990 Apr 26;322(17):1195-201. doi: 10.1056/NEJM199004263221705. PMID 2325710
- [Background] Cohn K, Gottesman L, Brennan M. Adrenocortical carcinoma. Surgery. 1986 Dec;100(6):1170-7. PMID 3787475
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0203.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Adrenal Cortex Neoplasms: Aggressive cancer that starts in the adrenal gland located at the top of the kidneys.
  Axitinib : 5 mg tab orally twice a day with food every 28 days
Period: Overall Study
Arm/Group | Adrenal Cortex Neoplasms
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adrenal Cortex Neoplasms
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 53.89 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR) of Axitinib Administered Daily, in Patients With Recurrent, Metastatic, or Primary Unresectable Adrenocortical Cancer (ACC)
Description: Response was defined by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is a disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameter. Progressive disease (PD) is a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm (Note: the appearance of one or more new lesions is also considered progression). Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking s reference the smallest sum diameters while on study.
Time Frame: 2 years
Measure: Number; unit: Participants
Arm/Group | Adrenal Cortex Neoplasms
Number analyzed (Participants) | 13
Participants
  Complete Response | 0
  Partial Response | 0
  Progression | 13
  Stable Disease | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse events module.
Time Frame: 3/2/11 - 8/2/12
Measure: Number; unit: Participants
Arm/Group | Adrenal Cortex Neoplasms
Number analyzed (Participants) | 13
Participants | 13

ADVERSE EVENTS:
Arm/Group | Adrenal Cortex Neoplasms
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adrenal Cortex Neoplasms (N=13)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adrenal Cortex Neoplasms (N=13)
Abdominal pain (Gastrointestinal disorders) | 6 (10)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (5)
Alkaline phosphatase increased (Investigations) | 5 (8)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (14)
Anorexia (Metabolism and nutrition disorders) | 4 (10)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (10)
Autoimmune disorder (Immune system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Blood bilirubin increased (Investigations) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
CPK increased (Investigations) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine increased (Investigations) | 4 (7)
Cushingoid (Endocrine disorders) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (9)
Dizziness (Nervous system disorders) | 2 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 7 (13)
Fever (General disorders) | 2 (2)
Gait disturbance (General disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 7 (7)
Hypertension (Vascular disorders) | 12 (76)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (13)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 3 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (6)
Hypothyroidism (Endocrine disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Lipase increased (Investigations) | 2 (6)
Lymphocyte count decreased (Investigations) | 6 (10)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (5)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Social circumstances - Other (auto accident) (Social circumstances) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Upper respiratory infection (Infections and infestations) | 2 (3)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight loss (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No